CLINICAL TRIAL: NCT04548050
Title: Impact of the Training of Nursing Staff on the Practice of Manual Expression of Early Colostrum in Neonatal Medicine
Acronym: ORLIKID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/CHU/26
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Early Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mothers informed by untrained nurse
- mothers informed by trained nurse
  Interventions: Other: Nurses training
- mothers informed by nurses trained 6 months ago
  Interventions: Other: Nurses training

INTERVENTIONS:
Other: Nurses training — * Presentation of the benefits of colostrum and manual expression technique on a slide show and practical workshops for learning the manual expression technique on a fictitious breast.
  * Presentation to all staff of a service protocol for early colostrum donation.
  Groups: mothers informed by nurses trained 6 months ago; mothers informed by trained nurse

SUMMARY:
Colostrum is an irreplaceable nutrient rich in protein and antibodies. Its taste and smell are similar to those of amniotic fluid (therefore rich for the senses of the baby separated from his mother). It should be offered to every newborn baby, regardless of term and the type of breastfeeding their mom wants. The early expression of colostrum, within the first 2 hours after childbirth, is an essential way to start lactation of a mother separated from her baby. The sooner and more often the mother stimulates her breasts, the more milk she will have for her baby in the weeks to come. Manual expression of milk is therefore an essential gesture to initiate lactation, maintain it, and giving colostrum to babies as early as possible is beneficial. Two studies carried out in the neonatal medicine department of Felix Guyon Hospital in premature infants <33 week of amenorrhea (PRE'OLACT study in 2015-2016 by Dr RAJAOFERA and Diploma from university (DU) breastfeeding brief in 2018-2019 by Dr GRONDARD) found the same results: the desire for breastfeeding is 80% but manual expression of colostrum before H24 is only achieved by 30% of mothers and before H6 in only 6% of cases.

.

ELIGIBILITY:
Inclusion Criteria:

* All mothers, over 18 years of age, of newborns hospitalized in neonatal medicine at the University Hospital Center (CHU) - Félix GUYON Hospital during the study period.
* Expressed no opposition from mothers to their participation and to the use of their data

Exclusion Criteria:

* Outborn
* Mother not hospitalized in the maternity ward of Félix Guyon Hospital
* Prognosis for the child engaged in the first 24 hours
* Difficult oral comprehension
* Medical contraindication to breastfeeding
* Unseen mother <3D

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All mothers, over 18 years of age, of newborns hospitalized in neonatal medicine at the CHU - Félix GUYON .
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
104/5000 Percentage of mothers who expressed colostrum before 24hours | 24hours after childbirth

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de la Réunion, Saint-Denis, France